CLINICAL TRIAL: NCT06708949
Title: A Randomized Phase 2 Trial of Nivolumab, Relatlimab Plus Ipilimumab vs. Nivolumab Plus Ipilimumab in First-line Advanced Renal Cell Carcinoma (RCC)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1337; NCI-2025-01553 (Other: Clinical Trials Reporting Program (CTR)
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Renal Cell Carcinoma, Clear Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment with Nivolumab + Ipilimumab (Experimental): Participants will randonmized to study and treatment will be administered on an outpatient basis.
  Interventions: Drug: Drugs Nivolumab; Drug: Ipilimumab
- Treatment with Nivolumab + Relatlimab + Ipilimumab (Experimental): Participants will randonmized to study and treatment will be administered on an outpatient basis.
  Interventions: Drug: Ipilimumab; Drug: BMS-986213 (Relatlimab-Nivolumab FDC)

INTERVENTIONS:
Drug: Drugs Nivolumab — Given by IV Infusion
  Arms: Treatment with Nivolumab + Ipilimumab
Drug: Ipilimumab — Given by IV Infusion
Drug: BMS-986213 (Relatlimab-Nivolumab FDC) — Given by IV Infusion
  Arms: Treatment with Nivolumab + Relatlimab + Ipilimumab

SUMMARY:
This is a phase 2 stratified, randomized, multicenter, study investigating the efficacy of a triplet arm treating with nivolumab 480 mg every 4 weeks (Q4W), relatlimab 160 mg Q4W and ipilimumab 1 mg/kg every 8 weeks (Q8W) intravenous (IV) versus a doublet arm treating with nivolumab 480 mg Q3W and ipilimumab 1mg/kg Q3W IV in first-line advanced RCC.

DETAILED DESCRIPTION:
Primary Objectives:

To determine the safety and tolerability of nivolumab, relatlimab and ipilimumab in patients with untreated advanced RCC

• To assess the ORR of nivolumab, relatlimab and ipilimumab in patients with untreated advanced RCC

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide a signed and dated written informed consent.
2. ≥ 18 years of age
3. Confirmed diagnosis of RCC with a clear cell component
4. Stage IV metastatic renal cell carcinoma per American Joint Committee on Cancer
5. No prior systemic therapy for RCC. Prior neo/adjuvant systemic therapy is not allowed.
6. Karnofsky performance status ≥ 70%.
7. At least one measurable lesion as defined by RECIST 1.1 (Appendix 3)

   • A tumor lesion situated in a previously irradiated area is considered a measurable/target lesion only if subsequent disease progression has been documented in the lesion
8. Adequate organ function within 28 days prior to first dose of protocol-indicated treatment, including:

   * White blood cell (WBC) ≥ 2,000 /µL
   * Absolute neutrophil count (ANC) ≥ 1,500/µL
   * Platelets ≥ 100,000/µL
   * Serum creatinine < 1.5 x upper limit of normal (ULN) or creatinine clearance > 30 mL/min (measured or calculated by Cockroft-Gault formula)
   * Total bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who must have total bilirubin < 3.0 mg/dL)
   * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN
9. Women must not be breastfeeding while taking the study drug and for up to five months after the last dose of study drug
10. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours prior to receiving first dose of protocol-indicated treatment. An extension up to 72 hours prior to the start of study treatment is permissible in situations where results cannot be obtained within the standard 24-hour window.

    * "Women of childbearing potential" (WOCBP) is defined as any female who has experienced menarche who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or is not postmenopausal.
    * Menopause is defined clinically as 12 months of amenorrhea in a woman over 45 years of age in the absence of other biological or physiological causes.
    * If menopausal status is considered for the purpose of evaluating childbearing potential, women < 62 years of age must have a documented serum follicle stimulating hormone (FSH) level within laboratory reference range for postmenopausal women, in order to be considered postmenopausal and not of childbearing potential.
11. Women of childbearing potential (WOCBP) must agree to follow instructions for acceptable contraception Appendix 5 from the time of signing consent, and for 23 weeks after their last dose of protocol-indicated treatment.

Exclusion Criteria:

1. Prior systemic treatment for RCC of any type including neoadjuvant or adjuvant therapy is not allowed.
2. ≤ 28 days before first dose of protocol-indicated treatment:

   • Major surgery requiring general anesthesia.
3. ≤ 14 days before first dose of protocol-indicated treatment:

   * Radiosurgery or radiotherapy
   * Minor surgery. (Note: Placement of a vascular access device is not considered minor or major surgery)
   * Active infection requiring infusion treatment.
4. Any history of or current CNS metastases
5. Any condition requiring systemic treatment with either corticosteroids (> 10 mg/day prednisone or equivalent daily) or other immunosuppressive medications within 14 days prior to initiating protocol-indicated treatment.

   • In the absence of active autoimmune disease, subjects are permitted the use of corticosteroids with minimal systemic absorption (e.g. topical, ocular, intra-articular, intranasal, and inhalational) ≤ 10 mg/day prednisone or equivalent daily; and physiologic replacement doses of systemic corticosteroids ≤ 10 mg/day prednisone or equivalent daily (e.g. hormone replacement therapy needed in patients with hypophysitis)
6. Active, known or suspected autoimmune disease (see Appendix 1 for a comprehensive list of autoimmune diseases and immune deficiencies).

   • Subjects with type I diabetes mellitus; endocrine organ dysfunction (e.g., hypothyroidism) that are controlled and only requiring only hormone replacement; skin disorders such as vitiligo, psoriasis or alopecia not requiring systemic treatment; or conditions not expected by the investigator to recur in the absence of an external trigger are permitted to enroll.
7. Known psychiatric condition, social circumstance, or other medical condition reasonably judged by the investigator to unacceptably increase the risk of study participation; or to prohibit the understanding or rendering of informed consent or anticipated compliance with and interpretation of scheduled visits, treatment schedule, laboratory tests and other study requirements.
8. History of myocarditis, regardless of etiology
9. Troponin T (TnT) or I (TnI) > 2× institutional upper limit of normal (ULN)

   • Participants with TnT or TnI levels between > 1× to 2× ULN will be permitted if repeat levels within 24 hours are ≤ 1× ULN. If TnT or TnI levels are between > 1× to 2× ULN within 24 hours, the participant may undergo a cardiac evaluation and be considered for treatment, based on a favorable benefit/risk assessment by the Investigator.

   When repeat levels within 24 hours are not available, a repeat test should be conducted as soon as possible. If TnT or TnI repeat levels beyond 24 hours are < 2× ULN, the participant may undergo a cardiac evaluation and be considered for treatment, based on a favorable benefit/risk assessment by the Investigator.
10. Treatment with any live/attenuated vaccine within 30 days of first study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
Safety and Averse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Eric Jonasch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (3):
- United States (3):
  - Duke University Medical Center, Durham, North Carolina
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2025-02-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT06708949/ICF_000.pdf